CLINICAL TRIAL: NCT03587480
Title: Total Mesorectal Excision(TME) With Lateral Lymph Node Dissection Versus TME After Neoadjuvant Chemo-radiotherapy of Lower Rectal Cancer With Suspected Local Lymph Node Metastasis
Brief Title: Total Mesorectal Excision(TME) With Lateral Lymph Node Dissection Versus TME After Neoadjuvant Chemo-radiotherapy
Acronym: TELEPHOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Luo-20180624
Record Dates: First submitted 2018-06-28; First posted 2018-07-16 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-03

CONDITIONS: Rectal Neoplasm Malignant
Keywords: Low rectal cancer; Total Mesorectal Excision (TME); neoadjuvant Chemo-radiotherapy (nCRT); lateral lymph node dissection (LLND)
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TME+LLND group (Other): Total Mesorectal Excision plus Lateral Lymph Node Dissection for low rectal cancer with regional lymph node metastasis.
  Interventions: Procedure: TME+LLND
- TME+nCRT group (Other): Total Mesorectal Excision After Neoadjuvant Chemo-radiotherapy for low rectal cancer with regional lymph node metastasis.
  Interventions: Procedure: TME+nCRT

INTERVENTIONS:
Procedure: TME+LLND — patients in TME+LLND group receive Lateral Lymph Node Dissection (LLND) after Total Mesorectal Excision(TME)
  Arms: TME+LLND group
Procedure: TME+nCRT — patients in TME+nCRT group receive Neoadjuvant Chemo-radiotherapy (nCRT) before Total Mesorectal Excision(TME)
  Arms: TME+nCRT group

SUMMARY:
Treatment for Low rectal cancer, especially in patients with regional lymph node metastasis are quite different between Japanese guideline (JSCCR) and western countries' guideline (NCCN, ESMO). While Japanese scholars advocate total mesorectal excision (TME) plus lateral lymph node dissection (LLND), European and American scholars advocate TME alone after Neoadjuvant Chemo-radiotherapy (nCRT), without the need of LLND. Accordingly, this clinical trial is designed to directly compare the efficacy and safety of these two treatment strategies for low rectal cancer with regional lymph node metastasis. It will provide high-level clinical evidence for the treatment of low rectal cancer with suspected local lymph node metastasis

DETAILED DESCRIPTION:
There are significant differences between Japanese guidelines (JSCCR) and Western guidelines (NCCN, ESMO) in the treatment of low rectal cancer, especially in patients with regional lymph node metastasis. Japanese scholars advocated total meso rectal resection (TME) + Lateral lymph node dissection (LLND), However, European and American scholars advocate that only TME is used after new adjuvant chemo-radiation (nCRT), without LLND. Therefore, the purpose of this clinical trial was to directly compare the efficacy and safety of these two treatment strategies for low rectal cancer with regional lymph node metastasis. This will provide a high level of clinical evidence for the treatment of low rectal cancer with suspected local lymph node metastasis

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma(below the peritoneal reflection) Clinical stage Ⅲ
2. Tumor is capable of performing radical recession
3. No past history of chemotherapy, pelvic radiation of other cancers.
4. Written informed consent
5. Lower tumor margin is confirmed below the peritoneal reflection
6. Clinical state T(1-3)N(1-2)M0 is confirmed by the multiple disciplines team(MDT) including surgeons,diagnostic radiologist,radiation oncologist and medical oncologists base on MRI and endorectal ultrasound -

Exclusion Criteria:

1. Past history of other cancers
2. Multiple Primary Colorectal Cancers or Familial adenomatous polyposis(FAP)
3. Combine with inflammatory bowl disease(IBD)
4. Recurrence tumor or invade other organs
5. Combine with obstruction,perforation or bleeding which need emergency surgery.
6. Local tumor invade the external sphincter, levator ani muscle or adjacent organs
7. Participant join other clinical trials in 4 weeks.
8. American Society of Anesthesiologists(ASA) ≥Ⅳ and/or Eastern Cooperative Oncology Group(ECOG) ≤2
9. Pregnant or lactating patients
10. Severity infection before operation
11. Psychological disorder
12. Severe dysfunction of organs or other contraindications
13. Cardiac infarction within six months
14. Severe pulmonary emphysema and pulmonary fibrosis
15. Doctor's decision for exclusion
16. Operative findings:

Tumor invade other organs Lower tumor margin is above the peritoneal reflection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2025-05-24 (Estimated); Study Completion 2030-05-24 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | From date of operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  36 months after surgery

SECONDARY OUTCOMES:
Operative time | Operation day
  Operation day
Blood loss | Operation day
  in the perioperative period
Incidence of sexual dysfunction | 3 years
  From the date of operation until the date of complication,assessed up to 3 years
Incidence of urinary dysfunction | 3 years
  From the date of operation until the date of complication,assessed up to 3 years
Incidence of defecation dysfunction | 3 years
  From the date of operation until the date of complication,assessed up to 3 years
incidence of Postoperative complications | 3 months
  From the date of operation until the date of complication,assessed up to 3 months
overall survival | From the date of operation until the date of death,assessed up to 5 years
  60 months after surgery
3-year local recurrence rate | From date of operation until the date of local-recurrence (up to 3 years)
  36 months after surgery
5-year disease-free survival | From date of operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  60 months after surgery
the score of quality of life | 3 months after operation
  The study investigate the quality of life using the WHOQOL Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yanxin Luo, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito M, Kobayashi A, Fujita S, Mizusawa J, Kanemitsu Y, Kinugasa Y, Komori K, Ohue M, Ota M, Akazai Y, Shiozawa M, Yamaguchi T, Akasu T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Urinary dysfunction after rectal cancer surgery: Results from a randomized trial comparing mesorectal excision with and without lateral lymph node dissection for clinical stage II or III lower rectal cancer (Japan Clinical Oncology Group Study, JCOG0212). Eur J Surg Oncol. 2018 Apr;44(4):463-468. doi: 10.1016/j.ejso.2018.01.015. Epub 2018 Jan 17. PMID 29428473
- [Background] Deng Y, Chi P, Lan P, Wang L, Chen W, Cui L, Chen D, Cao J, Wei H, Peng X, Huang Z, Cai G, Zhao R, Huang Z, Xu L, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Zhou Z, Cai Y, Kang L, Huang M, Peng J, Ren D, Wang J. Modified FOLFOX6 With or Without Radiation Versus Fluorouracil and Leucovorin With Radiation in Neoadjuvant Treatment of Locally Advanced Rectal Cancer: Initial Results of the Chinese FOWARC Multicenter, Open-Label, Randomized Three-Arm Phase III Trial. J Clin Oncol. 2016 Sep 20;34(27):3300-7. doi: 10.1200/JCO.2016.66.6198. Epub 2016 Aug 1. PMID 27480145
- [Background] Qin Q, Ma T, Deng Y, Zheng J, Zhou Z, Wang H, Wang L, Wang J. Impact of Preoperative Radiotherapy on Anastomotic Leakage and Stenosis After Rectal Cancer Resection: Post Hoc Analysis of a Randomized Controlled Trial. Dis Colon Rectum. 2016 Oct;59(10):934-42. doi: 10.1097/DCR.0000000000000665. PMID 27602924
- [Background] Huang M, Lin J, Yu X, Chen S, Kang L, Deng Y, Zheng J, Luo Y, Wang L, Lan P, Wang J. Erectile and urinary function in men with rectal cancer treated by neoadjuvant chemoradiotherapy and neoadjuvant chemotherapy alone: a randomized trial report. Int J Colorectal Dis. 2016 Jul;31(7):1349-57. doi: 10.1007/s00384-016-2605-7. Epub 2016 Jun 6. PMID 27270480
- [Result] Shinagawa T, Tanaka T, Nozawa H, Emoto S, Murono K, Kaneko M, Sasaki K, Otani K, Nishikawa T, Hata K, Kawai K, Watanabe T. Comparison of the guidelines for colorectal cancer in Japan, the USA and Europe. Ann Gastroenterol Surg. 2017 Dec 19;2(1):6-12. doi: 10.1002/ags3.12047. eCollection 2018 Jan. PMID 29863118
- [Result] Fujita S, Akasu T, Mizusawa J, Saito N, Kinugasa Y, Kanemitsu Y, Ohue M, Fujii S, Shiozawa M, Yamaguchi T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Postoperative morbidity and mortality after mesorectal excision with and without lateral lymph node dissection for clinical stage II or stage III lower rectal cancer (JCOG0212): results from a multicentre, randomised controlled, non-inferiority trial. Lancet Oncol. 2012 Jun;13(6):616-21. doi: 10.1016/S1470-2045(12)70158-4. Epub 2012 May 15. PMID 22591948
- [Result] Fujita S, Mizusawa J, Kanemitsu Y, Ito M, Kinugasa Y, Komori K, Ohue M, Ota M, Akazai Y, Shiozawa M, Yamaguchi T, Bandou H, Katsumata K, Murata K, Akagi Y, Takiguchi N, Saida Y, Nakamura K, Fukuda H, Akasu T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Mesorectal Excision With or Without Lateral Lymph Node Dissection for Clinical Stage II/III Lower Rectal Cancer (JCOG0212): A Multicenter, Randomized Controlled, Noninferiority Trial. Ann Surg. 2017 Aug;266(2):201-207. doi: 10.1097/SLA.0000000000002212. PMID 28288057
- [Result] Nagawa H, Muto T, Sunouchi K, Higuchi Y, Tsurita G, Watanabe T, Sawada T. Randomized, controlled trial of lateral node dissection vs. nerve-preserving resection in patients with rectal cancer after preoperative radiotherapy. Dis Colon Rectum. 2001 Sep;44(9):1274-80. doi: 10.1007/BF02234784. PMID 11584199
- [Result] Ogura A, Akiyoshi T, Nagasaki T, Konishi T, Fujimoto Y, Nagayama S, Fukunaga Y, Ueno M, Kuroyanagi H. Feasibility of Laparoscopic Total Mesorectal Excision with Extended Lateral Pelvic Lymph Node Dissection for Advanced Lower Rectal Cancer after Preoperative Chemoradiotherapy. World J Surg. 2017 Mar;41(3):868-875. doi: 10.1007/s00268-016-3762-0. PMID 27730352